CLINICAL TRIAL: NCT04957108
Title: Comparing Sensitivity and Specificity of Pacemaker ID Application and Cardiac Rhythm Management Device-Finder Application in Identifying Cardiac Implantable Electronic Device Manufacturer Using Chest Radiograph - an Observational Study.
Brief Title: Comparing Sensitivity and Specificity of Pacemaker ID Application and Cardiac Rhythm Management Device-Finder Application.
Status: Completed | Type: Observational
Sponsor: Aga Khan University Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Pirbhat Shams, Dr., Aga Khan University Hospital, Pakistan
Other Study IDs: 2020-5101-14156
Record Dates: First submitted 2021-06-22; First posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-06

CONDITIONS: Cardiac Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All cardiac implantable devices: Assessed separately by Pacemaker ID app and cardia-x algorithm
  Interventions: Other: Device identification using Xray.

INTERVENTIONS:
Other: Device identification using Xray. — PMIDa and CRMD-f applications were used to identify CIED

SUMMARY:
Smart phone-based applications to identify cardiac implantable electronic devices (CIED) are extremely useful in circumstances where urgent device interrogation is needed and device identification card is not available. Few studies have provided insight regarding the utility of these applications. We have studied two widely available applications i.e., Pacemaker ID app (PMIDa) or Cardiac Rhythm Management Devices-Finder (CRMD-f) to identiy device manufacturers in CIEDs.

DETAILED DESCRIPTION:
Smart phone-based applications to identify cardiac implantable electronic devices (CIED) are extremely useful in circumstances where urgent device interrogation is needed and device identification card is not available. Few studies have provided insight regarding the utility of these applications. We have studied two widely available applications i.e., Pacemaker ID app (PMIDa) or Cardiac Rhythm Management Devices-Finder (CRMD-f) to identiy device manufacturers in CIEDs.

547 patients who underwent CIED implantation from year 2016 - 2020 in our institute were enrolled. There were 438 Medtronic and 109 St. Jude's devices. All chest radiographs were de-identified and resized into 225*225 pixels focusing on the CIED. PMIDa and CRMD-f applications were used to identify CIED. Accuracy, sensitivity, specificity, negative predictive value, and positive predictive value for both applications were calculated and compared.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing CIED implantation and having xray post-implant at any point and time.

Exclusion Criteria:

* Patients with CIED for whome Xray was not available.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing CIED implantation and having post-device Xray were included.
Sampling Method: Non-Probability Sample
Enrollment: 547 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Accuracy sensitivity, specificity, negative predictive value, and positive predictive value for both Pacemaker ID app and CRMD finder app. | Upto 6 months of enrollment
  Accuracy, sensitivity, specificity, negative predictive value, and positive predictive value for both Pacemaker ID app and CRMD finder app. Above mentioned values shall be calculated after analysing data in SPSS and doing cross tabulation. Values will be in percentages.

SECONDARY OUTCOMES:
sensitivity, specificity, negative predictive value, and positive predictive value for both Pacemaker ID app and CRMD finder app. | Upto 6 months of enrollment
  sensitivity, specificity, negative predictive value, and positive predictive value for both Pacemaker ID app and CRMD finder app. Above mentioned values shall be calculated after analysing data in SPSS and doing cross tabulation. Values will be in percentages.

CONTACTS AND LOCATIONS:
Overall Officials: Yawer Saeed, MBBS, PHD, Principal Investigator — The Aga Khan University Hospital
Locations (1):
- The Aga Khan University, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: No